CLINICAL TRIAL: NCT05999877
Title: Non-interventional Cohort Study of Patients Previously Untreated or First-generation BTKi Intolerant With Chronic Lymphocytic Leukemia Describing the First-line Use of Acalabrutinib and Its Real-world Outcomes in Spain: the PICAROS Study
Brief Title: PICAROS - Acalabrutinib RWE on 1L CLL in Spain
Acronym: PICAROS
Status: Active, not recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D8221R00003
Record Dates: First submitted 2023-06-29; First posted 2023-08-21 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Observational; Chronic lymphocytic leukemia; Acalabrutinib
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a multicenter non-interventional study (NIS) on patients with CLL who have been treated with acalabrutinib for the first time within the year before the first site initiation visit in Spain

DETAILED DESCRIPTION:
This is a multicenter, non-interventional study (NIS) based on ambispective (including retrospective and/or prospective) real-world data collection of patients with CLL who have been treated with acalabrutinib for the first time within the year before the first site initiation visit, from approximately 50 Hospitals in Spain. Patients who had already initiated acalabrutinib therapy will be identified by the investigators and offered to participate in the study.

The start of acalabrutinib treatment (index date) must be prior to the first site initiation visit. Therefore, the clinical decision of starting patient on acalabrutinib has independently occurred prior to the patient inclusion into this study. Patients' eligibility for study inclusion is regardless of their current status of acalabrutinib therapy, for example, patients already deceased or discontinued therapy are still eligible to be included into this study. Patient data will be collected both retrospectively and/or prospectively up to 3.5 years from the first site initiation visit. For patients who received acalabrutinib therapy and have deceased, only retrospective medical chart review will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old at starting acalabrutinib treatment.
* Diagnosis of CLL.
* Start of acalabrutinib treatment (index date) in treatment-naïve CLL patients or those switching in first-line between first-generation BTK inhibitor to acalabrutinib due to intolerance in absence of progression according to routine clinical practice within the year before the first site initiation visit. Decision to administer acalabrutinib must be made and documented prior to inclusion into the study and must follow local clinical practice.
* Informed consent (for alive patients).

Exclusion Criteria:

* Enrolled in any clinical trial during acalabrutinib treatment.
* Patients who are unable to understand the study and its questionnaires due to insufficient knowledge of the Spanish language or their health status.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study aims to include approximately 315 patients who started acalabrutinib for the first time for the treatment of their CLL. They may include patients receiving acalabrutinib either as first treatment for their previously untreated CLL or patients who switched from first generation BTK inhibitor, used in first-line, to acalabrutinib due to intolerance.
  To minimize selection biases, all patients (alive or deceased) identified on acalabrutinib will be eligible for inclusion into the study.
  These patients will be included from approximately 50 hospitals distributed throughout Spain. The identification of patients for inclusion will be consecutive backwards until reaching a maximum of 15 patients per site.
Sampling Method: Non-Probability Sample
Enrollment: 192 (Actual)
Dates: Start 2023-07-11 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients on acalabrutinib therapy at 24 months after treatment initiation. | 24 months after treatment initiation.
  Proportion of patients on acalabrutinib therapy at 24 months after treatment initiation.
  In addition to this outcome measured in the overall population, it will also be assessed by the following factors:
  1. the reason for treatment initiation (i.e., first-line treatment-naïve patients, and those switching due to intolerance in absence of progression),
  2. presence/absence of risk factors (i.e., del17p, TP53 mutation, and unmutated IGHV).
  3. cardiovascular comorbidities (yes/no).

SECONDARY OUTCOMES:
Start dose in mg. | At acalabrutinib start date
  Acalabrutinib dose at starting treatment, overall and by the reason for treatment initiation (i.e., first-line treatment-naïve patients, and those switching due to intolerance in absence of progression).
Patients with acalabrutinib dose reductions (n, %), temporary interruptions (n, %), and permanent discontinuations (n, %). | From acalabrutinib start to acalabrutinib end, assessed up to 3.5 years of prospective study follow-up.
  Acalabrutinib dose reductions, temporary interruptions, and permanent discontinuations, overall and by the reason for treatment initiation (i.e., first-line treatment-naïve patients, and those switching due to intolerance in absence of progression).
Treatment duration in months. | From acalabrutinib start to acalabrutinib end, assessed up to 3.5 years of prospective study follow-up.
  Treatment duration, overall and by the reason for treatment initiation (i.e., first-line treatment-naïve patients, and those switching due to intolerance in absence of progression).
  Baseline patient characteristics associated with treatment duration in multivariate analyses, overall and according to the reason for treatment initiation (i.e., first-line treatment-naïve patients, and those switching due to intolerance in absence of progression).
Treatment adherence according to the percentage of days covered (PDC) while receiving acalabrutinib. | From acalabrutinib start to acalabrutinib end, assessed up to 3.5 years of prospective study follow-up.
  Treatment adherence according to the percentage of days covered (PDC) while receiving acalabrutinib, overall and by the reason for treatment initiation (i.e., first-line treatment-naïve patients, and those switching due to intolerance in absence of progression).
  The PDC will be based on data available on acalabrutinib treatment in pharmacy records, and defined as the percentage of days a patient has the medication available in a given period of time:
  PDC (%)=(No.days covered)/(No.days of interest)×100
TTNT (i.e., the time from the date of first dose of acalabrutinib to the first dose of the next treatment for CLL, or death from any cause [i.e. deaths are not censored]). | From the date of first dose of acalabrutinib to the first dose of the next treatment for CLL or death from any cause, whichever came first, assessed up to 3.5 years of prospective study follow-up.
  TTNT (i.e., the time from the date of first dose of acalabrutinib to the first dose of the next treatment for CLL, or death from any cause [i.e. deaths are not censored]), overall and according to the reason for treatment initiation (i.e., first-line treatment-naïve patients, and those switching due to intolerance in absence of progression).
OS (i.e., the time from the date of first dose of acalabrutinib to death from any cause). | From the date of first dose of acalabrutinib to death from any cause, whichever came first, assessed up to 3.5 years of prospective study follow-up.
  OS (i.e., the time from the date of first dose of acalabrutinib to death from any cause), overall and according to the reason for treatment initiation (i.e., first-line treatment-naïve patients, and those switching due to intolerance in absence of progression).
Adverse events that lead to acalabrutinib dose changes, temporary interruptions, or permanent discontinuation. Adverse events that are considered serious during acalabrutinib treatment. Events of clinical interest. | From acalabrutinib start to acalabrutinib end, assessed up to 3.5 years of prospective study follow-up.
  Adverse events that lead to acalabrutinib dose changes, temporary interruptions, or permanent discontinuation.
  Adverse events that are considered serious (including fatal events) during acalabrutinib treatment, globally and treatment related (when available).
  Events of clinical interest (atrial fibrillation, hypertension, bleeding, infections, ventricular arrhythmias, hepatotoxicity, secondary primary malignancies, cytopenia, and pneumonitis) during acalabrutinib treatment, globally and treatment related (when available).They will be described overall and according to the reason for treatment initiation (i.e., first-line treatment-naïve patients, and those switching due to intolerance in absence of progression).

OTHER OUTCOMES:
Best ORR (i.e., the proportion of patients that achieved complete or partial response) during acalabrutinib treatment. | From acalabrutinib start to acalabrutinib end, assessed up to 3.5 years of prospective study follow-up.
  Best ORR (i.e., the proportion of patients that achieved complete or partial response) during acalabrutinib treatment, overall and according to the reason for treatment initiation (i.e., first-line treatment-naïve patients, and those switching due to intolerance in absence of progression).
rwPFS (i.e., the time from the date of first dose of acalabrutinib to disease progression, or death from any cause). | From the date of first dose of acalabrutinib to disease progression or death from any cause, whichever came first, assessed up to 3.5 years of prospective study follow-up.
  rwPFS (i.e., the time from the date of first dose of acalabrutinib to disease progression, or death from any cause), overall and according to the reason for treatment initiation (i.e., first-line treatment-naïve patients, and those switching due to intolerance in absence of progression).
Scores on the EORTC QLQ-C30, its specific module for CLL QLQ-CLL17, and SATMED-Q during acalabrutinib treatment. | Study inclusion, month 3, month 6 and subsequent every 6 months during acalabrutinib treatment up to 3.5 years of prospective study follow-up.
  Scores on the EORTC Core Quality of Life questionnaire (EORTC QLQ-C30) and its specific module for CLL QLQ-CLL17 reported at inclusion, month 3, month 6 and subsequent every 6-month follow-up during acalabrutinib treatment.
  Satisfaction with acalabrutinib treatment reported at study inclusion, month 3, month 6 and subsequent every 6-month follow-up during acalabrutinib treatment (Treatment Satisfaction Questionnaire; SATMED-Q).
  These outcomes will be evaluated overall and according to the reason for treatment initiation (i.e., first-line treatment-naïve patients, and those switching due to intolerance in absence of progression).
Frequency of patients switching from capsules to tablets (if available). | From acalabrutinib start to acalabrutinib end, assessed up to 3.5 years of prospective study follow-up.
  Frequency of patients switching from capsules to tablets (if available).
Patient satisfaction after switching from capsules to tablets (if available). | From acalabrutinib start to acalabrutinib end, assessed up to 3.5 years of prospective study follow-up.
  Patient satisfaction according to SATMED-Q scores after switching from capsules to tablets (if available).
Patient adherence after switching from capsules to tablets (if available). | From acalabrutinib start to acalabrutinib end, assessed up to 3.5 years of prospective study follow-up.
  Patient adherence according to PDC after switching from capsules to tablets (if available).

CONTACTS AND LOCATIONS:
Locations (32):
- Spain (32):
  - Research Site, Almería, Andalusia
  - Research Site, Córdoba, Andalusia
  - Research Site, Granada, Andalusia
  - Research Site, Jaén, Andalusia
  - Research Site, Marbella, Andalusia
  - Research Site, Málaga, Andalusia
  - Research Site, Seville, Andalusia
  - Research Site, Zaragoza, Aragon
  - Research Site, Palma de Mallorca, Balearic Islands
  - Research Site, Las Palmas de Gran Canaria, Canary Islands
  - Research Site, San Cristóbal de La Laguna, Canary Islands
  - Research Site, Santander, Cantabria
  - Research Site, Salamanca, Castille and León
  - Research Site, Segovia, Castille and León
  - Research Site, Valladolid, Castille and León
  - Research Site, Guadalajara, Castille-La Mancha
  - Research Site, Toledo, Castille-La Mancha
  - Research Site, Barcelona, Catalonia
  - Research Site, Granollers, Catalonia
  - Research Site, L'Hospitalet de Llobregat, Catalonia
  - Research Site, Lleida, Catalonia
  - Research Site, Terrassa, Catalonia
  - Research Site, Ourense, Galicia
  - Research Site, Santiago de Compostela, Galicia
  - Research Site, Vigo, Galicia
  - Research Site, Madrid, Madrid
  - Research Site, Majadahonda, Madrid
  - Research Site, El Palmar, Murcia
  - Research Site, Murcia, Murcia
  - Research Site, Oviedo, Principality of Asturias
  - Research Site, Alicante, Valencia
  - Research Site, Valencia, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home